CLINICAL TRIAL: NCT04477785
Title: The Parkinson's Progression Markers Initiative (PPMI) Clinical - Establishing a Deeply Phenotyped PD Cohort
Brief Title: PPMI Clinical - Establishing a Deeply Phenotyped PD Cohort
Acronym: PPMI
Status: Recruiting | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Ken Marek, MD, Protocol Co- Principal Investigator, Institute for Neurodegenerative Disorders
Other Study IDs: PPMI-002
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson; Bio-markers; Neurodegenerative disorder; Imaging; Prodromal; Genetics; At Risk; Loss of Smell
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood will be obtained for the extraction of DNA to conduct sequencing and genomic analysis. These maybe collected in a fasted state.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical Observation: In PPMI Clinical up to 4,500 participants will be enrolled and followed longitudinally once identified, over the course of 5-8 years.

SUMMARY:
The Parkinson Progression Marker Initiative (PPMI) is a longitudinal, observational, multi-center natural history study to assess progression of clinical features, digital outcomes, and imaging, biologic and genetic markers of Parkinson's disease (PD) progression in study participants with manifest PD, prodromal PD, and healthy controls.

The overall goal of PPMI is to identify markers of disease progression for use in clinical trials of therapies to reduce progression of PD disability.

DETAILED DESCRIPTION:
PPMI is a broad program, expanding the goals of the original PPMI study, that includes this PPMI Clinical protocol, as well as other program initiatives such as the PPMI Remote, PPMI Digital App and PPMI Online protocols. Participants in PPMI may be asked to be enrolled in other PPMI program protocols, but depending on their method of recruitment, participants may be enrolled sequentially in varying order, as appropriate. PPMI participants may also be asked to participate in additional PPMI program initiatives (as they are developed), which may only involve a subset of PPMI participants based on their cohort designation and/or site location.

ELIGIBILITY:
7.1 Healthy Controls (HC) Note: Active Healthy controls previously enrolled in PPMI do not require re-assessment of eligibility criteria listed below for enrollment in PPMI Clinical. Active participants do need to be able to provide informed consent for PPMI Clinical participation (includes use of a designated research proxy).

7.1.1 Inclusion Criteria (HC)

1. Male or female age 57 years or older at Screening visit.
2. Individuals taking any of the following drugs: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, must be willing and medically able to hold the medication for at least 5 half-lives before SPECT imaging.
3. Confirmation that participant is eligible based on Screening SPECT imaging.
4. Able to provide informed consent.
5. Either is male, or is female and meets additional criteria below, as applicable:

   * Female of childbearing potential who is not pregnant, lactating, or planning pregnancy during the study and has a negative pregnancy test on day of Screening SPECT imaging test prior to injection of DaTscanTM.

7.1.2 Exclusion Criteria (HC)

1. First degree relative with PD (i.e., biologic parent, sibling, child).
2. Current or active clinically significant neurological disorder (in the opinion of the Investigator).
3. Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
4. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine within 6 months of Screening visit.
5. Current treatment with anticoagulants (e.g., coumadin, heparin, oral thrombin inhibitors) that might preclude safe completion of the lumbar puncture.
6. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
7. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
8. Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

7.2 Parkinson's Disease (PD) Note: Active PD participants previously enrolled in PPMI do not require re-assessment of eligibility criteria listed below for enrollment in PPMI Clinical. Active participants do need to be able to provide informed consent for PPMI Clinical participation (includes use of a designated research proxy).

7.2.1 Inclusion Criteria (PD)

1. Male or female age 30 years or older at Screening Visit.
2. A diagnosis of Parkinson's disease for 2 years or less at Screening Visit.
3. Not expected to require PD medication within at least 6 months from Baseline.
4. Patients must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia); OR either asymmetric resting tremor or asymmetric bradykinesia.
5. Hoehn and Yahr stage I or II at Baseline.
6. Individuals taking any of the following drugs: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, must be willing and medically able to hold the medication for at least 5 half-lives before SPECT imaging.
7. Confirmation that participant is eligible based on Screening SPECT imaging.
8. Able to provide informed consent.
9. Either is male, or is female and meets additional criteria below, as applicable:

   * Female of childbearing potential who is not pregnant, lactating, or planning pregnancy during the study and has a negative pregnancy test on day of Screening SPECT imaging test prior to injection of DaTscanTM.

7.2.2 Exclusion Criteria (PD)

1. Currently taking levodopa, dopamine agonists, MAO-B inhibitors, amantadine or another PD medication, except for low-dose treatment of restless leg syndrome (with permission of medical monitor).
2. Has taken levodopa, dopamine agonists, MAO-B inhibitors or amantadine within 60 days of Baseline visit.
3. Has taken levodopa or dopamine agonists prior to Baseline visit for more than a total of 90 days.
4. Atypical PD syndromes due to either drugs (e.g., metoclopramide, flunarizine, neuroleptics) or metabolic disorders (e.g., Wilson's disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy).
5. A clinical diagnosis of dementia as determined by the investigator.
6. Previously obtained MRI scan with evidence of clinically significant neurological disorder (in the opinion of the Investigator).
7. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine within 6 months of Screening visit.
8. Current treatment with anticoagulants (e.g., coumadin, heparin, oral thrombin inhibitors) that might preclude safe completion of the lumbar puncture.
9. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
10. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
11. Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

7.3 Parkinson's Disease (PD) with LRRK2 or GBA variant Note: Active PD participants previously enrolled in PPMI do not require re-assessment of eligibility criteria listed below for enrollment in PPMI Clinical. Active participants do need to be able to provide informed consent for PPMI Clinical participation (includes use of a designated research proxy).

7.3.1 Inclusion Criteria (PD ¬- LRRK2 or GBA)

1. Male or female age 30 years or older at Screening Visit.
2. A diagnosis of Parkinson's disease for 2 years or less at Screening Visit.
3. Patients must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia); OR either asymmetric resting tremor or asymmetric bradykinesia.
4. Hoehn and Yahr stage I or II at Baseline.
5. Confirmation of causative LRRK2 or GBA (willingness to undergo genetic testing as part of genetic screening and be informed of genetic testing results, or approved documentation of prior genetic testing results).
6. Individuals taking any of the following drugs: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, must be willing and medically able to hold the medication for at least 5 half-lives before SPECT imaging.
7. Confirmation that participant is eligible based on Screening SPECT imaging.
8. Able to provide informed consent.
9. Either is male, or is female and meets additional criteria below, as applicable:

   * Female of childbearing potential who is not pregnant, lactating, or planning pregnancy during the study and has a negative pregnancy test on day of Screening SPECT imaging test prior to injection of DaTscanTM.

7.3.2 Exclusion Criteria (PD - LRRK2 or GBA)

1. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine within 6 months of Screening visit.
2. Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
3. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
4. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
5. Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

7.4 Parkinson's Disease (PD) with SNCA or rare genetic variant Note: Active PD participants previously enrolled in PPMI do not require re-assessment of eligibility criteria listed below for enrollment in PPMI clinical. Active participants do need to be able to provide informed consent for PPMI Clinical participation (includes use of a designated research proxy).

7.4.1 Inclusion Criteria (PD - SNCA or rare genetic variant (such as Parkin or Pink1))

1. Male or female age 30 years or older at Screening Visit.
2. Parkinson's disease diagnosis at Screening Visit.
3. Patients must have at least two of the following: resting tremor, bradykinesia, rigidity (must have either resting tremor or bradykinesia); OR either asymmetric resting tremor or asymmetric bradykinesia.
4. Hoehn and Yahr stage I, II, or III at Baseline.
5. Confirmation of causative SNCA or rare genetic variant (such as Parkin or Pink1) (willingness to undergo genetic testing as part of genetic screening and be informed of genetic testing results, or approved documentation of prior genetic testing results).
6. Individuals taking any of the following drugs: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, must be willing and medically able to hold the medication for at least 5 half-lives before SPECT imaging.
7. Confirmation that participant is eligible based on Screening SPECT imaging.
8. Able to provide informed consent.
9. Either is male, or is female and meets additional criteria below, as applicable:

   * Female of childbearing potential who is not pregnant, lactating, or planning pregnancy during the study and has a negative pregnancy test on day of Screening SPECT imaging test prior to injection of DaTscanTM.

7.4.2 Exclusion Criteria (PD - SNCA or rare genetic variant (such as Parkin or Pink1))

1. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine within 6 months of Screening visit.
2. Current treatment with anticoagulants (e.g., coumadin, heparin) that might preclude safe completion of the lumbar puncture.
3. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
4. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
5. Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

7.5 Prodromal Note: Active Prodromal participants previously enrolled in PPMI do not require re-assessment of eligibility criteria listed below for enrollment in PPMI Clinical. Active participants do need to be able to provide informed consent for PPMI Clinical participation (includes use of a designated research proxy).

The specific predictive eligibility criteria for participants recruited through PPMI Remote to advance to PPMI Clinical will be iteratively optimized based on data collected from these studies.

7.5.1 Inclusion criteria (Prodromal)

For Screening:

1. Confirmation that participant is eligible based on centrally determined predictive criteria including the University of Pennsylvania Smell Identification Test (UPSIT).

   * For participants in PPMI Remote, referral to the clinical site confirms predictive eligibility.
   * For participants identified by the clinical site, predictive criteria are based on generalized risk such as first degree biologic relative, known risk of PD including RBD, or known genetic variants associated with PD risk.

   Additionally, confirmation of UPSIT eligibility during the Screening visit prior to SPECT Imaging.
2. Male or female age 60 years or older (except age 30 years or older for SNCA, or rare genetic variants (such as Parkin or Pink1) participants).
3. Individuals taking any of the following drugs: alpha methyldopa, methylphenidate, amphetamine derivatives or modafinil, must be willing and medically able to hold the medication for at least 5 half-lives before SPECT imaging.
4. Able to provide informed consent.
5. Either is male, or is female and meets additional criteria below, as applicable:

   • Female of childbearing potential who is not pregnant, lactating, or planning pregnancy during the study and has a negative pregnancy test on day of Screening SPECT imaging test prior to injection of DaTscanTM.

   For continuation to Baseline visit and ongoing follow-up:
6. Confirmation that participant is eligible based on *Screening SPECT imaging.

   * Screening SPECT Imaging eligibility:

Based on the results of the SPECT imaging test, Prodromal participants eligible to continue their participation in PPMI Clinical will be asked to return for their PPMI Clinical baseline visit. Neither the participant nor the site investigator will be made aware of the participant's DAT status during the study.

* It is anticipated that approximately 6,000 participants will complete a screening visit to undergo DAT imaging. Approximately 2,000 participants will be eligible to continue their participation in PPMI Clinical (those not eligible to proceed will remain in PPMI Remote, as applicable).
* All participants with DAT deficit will be eligible to continue their participation in PPMI Clinical. It is estimated that about 75% of eligible participants will have a DAT deficit (defined by a hybrid of visual assessment and quantitative striatal specific binding analysis).
* Some participants without DAT deficit will also be eligible to continue their participation in PPMI Clinical. These participants will be chosen based on DAT binding that is reduced from age expected but it not outside the normal range and/or from individuals with high-risk of PD including RBD, LRRK2, GBA, SNCA, or rare genetic variants (such as Parkin or Pink1) that do not demonstrate DAT deficit. It is estimated that about 25% of eligible participants will not have a DAT deficit.
* It is anticipated that approximately 30% of the PPMI Clinical prodromal participants with DAT deficit will phenoconvert to motor parkinsonism during a 3 to 5-year follow-up.

7.5.2 Exclusion Criteria (Prodromal)

1. Clinical diagnosis of PD at screening, other parkinsonism, or dementia.
2. Received any of the following drugs: dopamine receptor blockers (neuroleptics), metoclopramide and reserpine within 6 months of Baseline Visit.
3. Current treatment with anticoagulants (e.g. coumadin, heparin) that might preclude safe completion of the lumbar puncture.
4. Condition that precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
5. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.
6. Currently taking levodopa, dopamine agonists, MAO-B inhibitors, amantadine or another PD medication, except for low-dose treatment of restless leg syndrome (with permission of medical monitor).
7. Has taken levodopa, dopamine agonists, MAO-B inhibitors or amantadine within 60 days of Baseline visit. except for low-dose treatment of restless leg syndrome (with permission of medical monitor).
8. Any other reason that, in the opinion of the investigator, would render the participant unsuitable for study enrollment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In PPMI Clinical up to 4,500 participants will be enrolled and followed longitudinally from approximately 50-55 international clinical sites across a variety of cohorts, including healthy controls, Parkinson disease, PD manifesting gene carriers, and Prodromal (those at risk for developing PD).
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Establish standardized protocols for acquisition, transfer and analysis of clinical, digital, imaging, biologic and genetic data that can be used by the PD research community. | Baseline to 156 months
  This protocol will build on the existing PPMI infrastructure
Comprehensive and uniformly acquired dataset | Baseline to 156 months
  Develop a comprehensive and uniformly acquired clinical, digital and imaging dataset and repository of biological and genetic samples that would be available to the PD research community to test hypotheses of the underlying molecular pathobiology of PD, enable modeling of PD progression to identify clinical and/or data driven PD progression sub-sets, and inform studies testing PD therapeutics (for examples, clinical trials targeting synuclein, LRRK2, GBA as well as other targets)
Comparison between Rates of Change | Study intervals ranging from 3 months to 156 months
  Use clinical and biological data to estimate the mean rates of change and the variability around the mean of clinical, digital, imaging, biological and genetic outcomes in study participants with PD diagnosis (including patients with a LRRK2, GBA, SNCA or rare genetic variants (such as Parkin or Pink1) and individuals with prodromal Parkinson's disease (including individuals with REM sleep behavior disorder (RBD)), olfactory loss, LRRK2, GBA, SNCA or rare genetic variants (such as Parkin or Pink1) and/or other risk factors for PD with and without dopamine transporter (DAT) deficit and in healthy participants.
Prevalence of measures of clinical, imaging and biomic outcomes in various subsets | study intervals ranging from baseline to 156 months.
  Confirm existing and identify novel clinical, digital, imaging, biologic and genetic PD progression markers to identify quantitative individual measures or combinations of measures that demonstrate optimum interval change in study participants with PD diagnosis (including patients with a LRRK2, GBA, SNCA or rare genetic variants (such as Parkin or Pink1)) and individuals with prodromal Parkinson's disease (including individuals with RBD, olfactory loss, a LRRK2, GBA, SNCA or rare genetic variants (such as Parkin or Pink1) and/or other risk factors for PD with and without DAT deficit in comparison to healthy controls or in sub-sets of study participants with PD diagnosis or prodromal PD defined by baseline assessments, progression milestones and/or rate of clinical, digital, imaging, biologic and genetic change, or other measures.
Establish the probability of phenoconversion to PD | study intervals ranging from baseline to 156 months.
  Evaluate the probability of phenoconversion to PD for individuals with prodromal PD enrolled in the prodromal cohorts (including individuals with RBD, olfactory loss, a LRRK2, GBA, SNCA or rare genetic variants (such as Parkin or Pink1) and/ or other risk factors for PD with and without DAT deficit).

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth L Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders; Caroline Tanner, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (50):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Foundation for Medical Education and Research, Scottsdale, Arizona
  - Banner Research Institute, Sun City, Arizona
  - University of California San Diego, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Institute For Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease& Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - Beth Israel Medical Center, New York, New York
  - NYU Langone Health, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati/Cincinnati Children's Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health &Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Univ of Washington and VA Puget Sound Health Care System, Seattle, Washington
- Innsbruck Medical University, Innsbruck, Austria
- Canada (3):
  - The Ottawa Hospital - Civic Campus, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec
- Germany (4):
  - Philipps-University of Marburg, Hessen
  - Paracelsus-Elena Klinik, Kassel
  - University of Luebeck, Lübeck
  - University of Tuebingen, Tübingen
- Foundation for Biomedical Research of the Academy of Athens, Athens, Greece
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- University of Salerno, Salerno, Italy
- Parkinson Research Clinic, Luxembourg, Luxembourg
- Radboud University, Nijmegen, Gelderland, Netherlands
- Lagos College of Medicine, University of Lagos, Lagos, Nigeria
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian
- United Kingdom (4):
  - Queen Mary University of London, London, Britain
  - Newcastle University, Newcastle upon Tyne, Tyne and Wear
  - Imperial College London, London
  - John Radcliffe Hospital Oxford and Oxford University, Oxford

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pacheco Pachado M, Casas AI, Elbatreek MH, Nogales C, Guney E, Espay AJ, Schmidt HHHW. Re-Addressing Dementia by Network Medicine and Mechanism-Based Molecular Endotypes. J Alzheimers Dis. 2023;96(1):47-56. doi: 10.3233/JAD-230694. PMID 37742653